CLINICAL TRIAL: NCT05964153
Title: Pilot Study of Liquid Biopsy as a Diagnostic Tool for Gliomas by Analyzing Circulating Tumor DNA in Blood Samples, and Its Validation With the Corresponding Tissue Biopsies.
Brief Title: Analysis of Circulating DNA in Blood Samples of Glioma-affected Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Silvia Gil-Duran, Principal Investigator, Corporacion Parc Tauli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: I3PT_SG2022_01
Record Dates: First submitted 2023-04-04; First posted 2023-07-27 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Glioma; Circulating Tumor Cell
Keywords: Liquid Biopsy; Glioma; Circulating free DNA; ddPCR
MeSH Terms: conditions — Glioma; Neoplastic Cells, Circulating | interventions — Liquid Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Circulating free DNA analysis (Experimental): * Correlate the results of the tissue samples with those of the blood samples, the concentration of ctDNA found, and the magnetic resonance images prior to the biopsies.
  * Compare other variables such as time, money, and the impact on the patient (recovery time after biopsies, pain, sequelae,...) between the liquid biopsy procedure and the conventional tissue biopsy procedure.
  Interventions: Diagnostic Test: Liquid Biopsy

INTERVENTIONS:
Diagnostic Test: Liquid Biopsy — Analysis of the circulating free DNA in blood patients affected by gliomas

SUMMARY:
The present pilot study aims to investigate a new strategy in the liquid biopsy protocol for the diagnosis of gliomas based on the detection of circulating tumor DNA in the blood of patients with brain lesions compatible with this type of tumor.

In order to increase the sensitivity of the technique, the investigators will work with raw blood samples through minimally invasive procedures. The subsequent analysis will be done with digital PCR, due to its low detection limit. The mutational results of each patient's samples will be compared with those obtained from the corresponding tissue biopsies. This step will allow the team to determine the robustness and reliability of the liquid biopsy. The grading of the tumor, as well as the confirmation of the diagnosis, will be obtained from the histological data.

With the inclusion of more patients in the future, and with the optimization of the mutations investigated, the investigators want to standardize the protocol for the diagnosis of gliomas with liquid biopsy. This technique is less invasive than current surgical procedures used for diagnosis. In addition, using fewer hospital resources should allow a more accurate and rapid diagnosis of the pathology, and therefore, start the more personalized therapeutic stage earlier.

DETAILED DESCRIPTION:
Currently, brain tumors are detected by means of an imaging technique (usually magnetic resonance imaging) with a contrast agent. The determination of the type of tumor, as well as its grading, is usually done subsequently with a biopsy of the tissue, where different solid samples are extracted as representative as possible to analyze them in the Pathological Anatomy service. Nevertheless, there are some factors that limit surgical access, such as: the advanced age of the patient, the location of the tumor in eloquent or risky areas, as well as the presence of large tumors with very diffuse borders. In these cases, the diagnosis of the brain tumor is usually made directly with the magnetic resonance image, which implies a risk of error due to the lack of clinical information from this test.

Limitations like these make the minimally invasive procedure of liquid biopsy an extremely necessary diagnostic tool. For this reason, the investigators want to start a pilot study of this technique in those patients with brain lesions in the resonance images compatible with a glioma-like tumor.

In particular, the main aim of the study is to analyze the blood samples obtained from these patients in order to detect and quantify the circulating DNA (ctDNA) of tumor cells on it. These DNA fragments are expelled into the bloodstream by mechanisms still unknown as a result of numerous processes of apoptosis and necrosis of tumor cells. By analyzing them through a ddPCR, the investigators will try to detect the specific mutations present in this tumoral ctDNA, allowing the team to confirm the presence of a glioma-type tumor, and providing real-time information of its classification as astrocytoma or oligodendroglioma.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* De novo primary brain lesion, compatible with a glioma according to contrast-enhanced magnetic resonance images. The injury must be treated by the usual surgical procedure.
* Signature of informed consent.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Reasonable doubts in the diagnosis of glioma by magnetic resonance, or patients whose tissue biopsy diagnoses a brain lesion other than a glioma.
* Patients who cannot undergo surgical resection, or when the tissue samples taken are not significant enough to be analyzed.
* Inability or disagreement with signing the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Circulating free DNA detection | 1 year (2023-2024)
  Circulating free DNA detection in blood samples of patients by means of a ddPCR

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Gil, Principal Investigator — Hospital Universitari Parc Taulí
Locations (1):
- Hospital Universitari Parc Taulí, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No